CLINICAL TRIAL: NCT05293470
Title: A Post Marketing Surveillance on Piqray (Alpelisib) in Korea
Brief Title: A Post Marketing Surveillance on Piqray in Korea
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719CKR01
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; NIS; Piqray; Korea; Alpelisib
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Piqray: Patients prescribed with Piqray
  Interventions: Other: Piqray

INTERVENTIONS:
Other: Piqray — There is no treatment allocation. Patients administered Piqray by prescription will be enrolled.
  Other Names: Alpelisib

SUMMARY:
This is a prospective, multicenter, open-label, non-comparative, non-interventional, observational study to assess te safety and effectiveness of Piqray in the real-world setting

DETAILED DESCRIPTION:
The observation duration will be up to 24 weeks after enrollment, which is sufficient to provide adequate information about the safety and effectiveness of Piqray. If the subject does not return for a follow-up visit or stops taking Piqray for any reason, all data collected until the date of the last contact of the subject will be used. Patients will be followed up (safety follow up) for 30 days afetr either 24 weeks-treatment or early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this study must meet all of the following criteria:

1. Postmenopausal women and men who have a confirmed diagnosis of hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative, PIK3CA mutated, advanced or metastatic breast cancer.
2. Patients who have progressed on prior endocrine based therapy and are going to start Piqray treatment for the first time in accordance with the locally approved label.
3. Patients who are willing to provide written informed consent

Exclusion Criteria:

Subjects eligible for this study must not meet the following criteria:

1. Patients with contraindication according to prescribing information for Piqray in Korea.

   - Severe hypersensitivity to Piqray or to any of its components
2. Female subjects who are pregnant and nursing (lactating)
3. Patients who are sexually active but not willing to follow contraceptive precautions during taking Piqray.
4. Participants who receive or are going to receive any investigational medicine during surveillance period.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are going to receive Piqray per locally approved label are eligible and will be prescribed with Piqray under routine medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | 24 weeks
  Incidence of AEs, including SAEs and ADRs

SECONDARY OUTCOMES:
Objective response rates (ORRs) | Up to 24 weeks
  Objective response rates (ORRs). ORR is defined as the proportion of treated patients who achieve a best overall response (BOR) of partial response (PR) or complete response (CR) according to the response evaluation criteria in solid tumors (RECIST) version 1.1.
Prescription dose of Piqray in combination with fulvestrant | Up to 24 weeks
  Prescription dose of Piqray in combination with fulvestrant

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- South Korea (10):
  - Novartis Investigative Site, Cheonan Si, Chungcheongnam-do
  - Novartis Investigative Site, Daegu, Dalseo gu
  - Novartis Investigative Site, Deogyang Gu Goyang Si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Jeollanam
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No